CLINICAL TRIAL: NCT01022385
Title: The Effect of a Very Low-residual Diet on the Preparation Before Capsule Endoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Dr. Eva Niv, Hillel Yaffe Medical Center
Purpose: Diagnostic
Other Study IDs: 0064-08-HYMC
Record Dates: First submitted 2009-11-26; First posted 2009-12-01 (Estimated); Last update posted 2009-12-01 (Estimated); Status verified 2009-11

CONDITIONS: Gastrointestinal Complaints

ARMS (2):
- 12-hour fast (No Intervention)
- 24-hour low-residual diet and 12-hour fast (Active Comparator)
  Interventions: Dietary Supplement: 24-hour low-residual diet

INTERVENTIONS:
Dietary Supplement: 24-hour low-residual diet
  Arms: 24-hour low-residual diet and 12-hour fast

SUMMARY:
The aim of the proposed study is to compare prospectively two methods of small bowel preparation prior capsule endoscopy study, the effect on the cleanliness and the quality of visualization after two protocols of preparation: a 12 hour fast only versus 24 hour of a very low residual diet (ENSURE, Abbott Laboratories, Israel) + 12 hour fast.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients who will submitted to capsule endoscopy due to following medical indications:

  * suspected Crohn's disease
  * obscure GI bleeding
  * iron deficiency anemia
  * suspected malabsorption disease
  * unexplained abdominal pain
  * unexplained chronic diarrhea

Exclusion Criteria:

* pregnancy
* patients who had previous surgery on Gastrointestinal tract
* patients with previous intestinal obstruction
* patients who will refuse to participate in the study
* diabetes mellitus
* known celiac disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2009-12; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Cleanliness and better visualization of the small bowel during capsule endoscopy | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel